CLINICAL TRIAL: NCT01518426
Title: Evaluation of Evoked Potentials Recording Modalities in Healthy Volunteer Population.
Acronym: 3Electrods
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-A00102-39
Record Dates: First submitted 2011-12-22; First posted 2012-01-26 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Attitude to Computers
Keywords: Brain computer interface; EEG recording; Electrodes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Extraction of P300 ERPs (Experimental): Extract P300 ERPs with Emotiv EEG headset
  Interventions: Device: EEG Recording (Emotiv)

INTERVENTIONS:
Device: EEG Recording (Emotiv) — Record EEG during auditory oddball paradigms:
  * with Emotiv EEG headset EMOTIV CAP (see http://www.emotiv.com)
  * with 3 electrodes : 3 different types of electrodes at the time (needle, cupule 5mm, cupule 10mm)
  Other Names: EEG recording

SUMMARY:
The purpose of this study is to compare three different techniques of EEG recording for extraction of P300 Evoked Related Potentials (ERPs).

DETAILED DESCRIPTION:
Brain Computer Interface (BCI) are used to restore control and communication in patient with severe disabilities such as Locked In Syndrome (LIS) patients.

The aim of this study is to identify the most relevant recording technique for extraction of P300 ERPs in EEG signals. Three different electrodes (needle, standard ,silver) will be simultaneously compared in a prospective design in 10 healthy volunteers, as suggested by principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers male or female aging over 18
* Signed informed consent
* Passed the preliminary exam
* Registered in the national database for persons willing to participate in Biomedical research

Exclusion Criteria:

* Visual or hearing problems
* Cognitive problems
* Illiterate persons
* Persons under Guardianship or Trusteeship
* Having Epilepsy
* Pregnant women Not covered by the social security system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Wilcoxon statistic (Area Under the Curve) | T0+2h (end of each technique)
  An Linear Discriminant Analysis (LDA) will be used to discriminate target and Algorithm performance (Wilcoxon statistic) for discrimination between occurrent and non-occurrent stimuli.
  Signals will adequately be pre-processed: denoised and spatialy filtered (xDAWN). The Area Under the Receiver Operator Characteristic Curve (AUC) also called wilcoxon statistic will be used to identify the signals of best quality.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Mayaud, ENGINEER, Study Director — Centre d'Investigation Clinique et Technologique 805
Locations (1):
- Raymond Poincaré Hospital, Garches, Paris Area, France